CLINICAL TRIAL: NCT06038591
Title: Parenting Intervention to Improve Young Children's Sleep Among Families With Low Income
Brief Title: Parent Intervention to Improve Child Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Temple University (Other); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Elizabeth Adams, Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00123879; 5P20GM130420 (NIH)
Record Dates: First submitted 2023-08-28; First posted 2023-09-15 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Sleep

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sleep Intervention (Experimental): The sleep intervention focuses on enhancing young children's sleep by providing parents with behavioral strategies and support. Interventionists will work with parents on establishing consistent soothing bedtime routines; behavioral regulation to manage bedtime resistance and nighttime wakings; goal setting, problem solving, and action planning; self-monitoring via daily sleep logs; and stimulus control of child's sleep environment.
  Interventions: Behavioral: Sleep Tight
- Comparison/control (No Intervention): The comparison arm is a no-contact control group. Parents and children will not receive any intervention. They will be placed on a wait-list, and then offered the sleep intervention once the post-assessments are complete.

INTERVENTIONS:
Behavioral: Sleep Tight — The sleep intervention focuses on enhancing young children's sleep by providing parents with behavioral strategies and support. Interventionists will work with parents on establishing consistent soothing bedtime routines; behavioral regulation to manage bedtime resistance and nighttime wakings; goal setting, problem solving, and action planning; self-monitoring via daily sleep logs; and stimulus control of child's sleep environment.
  Arms: Sleep Intervention

SUMMARY:
In this study, the investigators pilot tested a parenting intervention to improve young children's sleep in families with low income. Families were randomized to an intervention or wait-list control group. The investigators hypothesized the intervention would be feasible and acceptable to enrolled families.

DETAILED DESCRIPTION:
This pilot study tested a parenting intervention to improve young children's sleep in families with low income using a randomized controlled trial (RCT) design. Parents were randomized to the intervention or wait-list control group. Intervention content was delivered in virtual sessions with a parent and interventionist. The primary aim was to examine intervention feasibility (e.g., recruitment, retention, acceptability) with a secondary goal of preliminary efficacy on intervention changes in child sleep patterns to inform a future large-scale RCT. Exploratory evidence was collected on changes in children's health behaviors (e.g., diet, screen time), and social-emotional health (e.g., behavior problems) as indicators for potential spillover effects on these domains.

ELIGIBILITY:
Inclusion Criteria:

* Parents or primary caregivers 18 years of age or older
* Have a child 2-4 years of age
* Child's 24-hour sleep duration does not meet established recommendations based on child age
* English speaking
* Annual household income <= 200% of the Federal Poverty Line or receive assistance benefits (e.g., SNAP, WIC)
* Computer or phone access for video calls

Exclusion Criteria:

* Parent or child has a medical condition that impairs their ability to participate
* Child has a clinical sleep disorder
* Child takes medication that significantly impacts their sleep

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Intervention feasibility: recruitment screening eligibility | Through study completion, an average of 2 years
  Percent of children screened who were eligible
Intervention feasibility: recruitment screening enrollment | Through study completion, an average of 2 years
  Percent of eligible children who were enrolled
Intervention feasibility: recruitment duration | Through study completion, an average of 2 years
  Duration to reach the target sample
Intervention feasibility: Enrollment yield for each recruitment strategy | Through study completion, an average of 2 years
  Percent of enrolled participants that were recruited via each recruitment strategy to determine the highest and lowest yielding strategies.
Intervention feasibility: retention attendance | Through study completion, an average of 2 years
  Percent attendance at assessment visits
Intervention feasibility: retention percentage | Through study completion, an average of 2 years
  Percent of sample retained at post-intervention
Intervention feasibility: retention dropout | Through study completion, an average of 2 years
  Percent of sample that drops out or is lost to follow-up
Intervention feasibility: retention dropout reasons | Through study completion, an average of 2 years
  Reasons for dropping out of the study
Intervention acceptability | Through study completion, an average of 2 years
  Acceptability will be assessed in an exit survey with Likert scale items and open-ended questions about intervention likes/dislikes and suggestions for future changes. Likert scale values range 1-5. Higher numbers indicate better outcomes (e.g., more positive acceptability)

SECONDARY OUTCOMES:
Process measures: Intervention attendance | Through study completion, an average of 2 years
  Proportion of intervention sessions attended, including makeup sessions, obtained from attendance records.
Process measures: Content fidelity | Through study completion, an average of 2 years
  Checklist completed by researchers for each intervention session that evaluates the extent to which the program content was addressed
Process measure: Implementation | Through study completion, an average of 2 years
  Survey checklist completed by interventionists after each intervention session that assess implementation barriers
Child sleep: night sleep duration | Baseline (0 weeks) and post-intervention (6 weeks)
  Wrist-worn actigraphy devices were used to calculate child's nighttime sleep duration
Child sleep: daytime sleep duration | Baseline (0 weeks) and post-intervention (6 weeks)
  Wrist-worn actigraphy devices were used to calculate child's daytime sleep duration
Child sleep: 24-hour sleep duration | Baseline (0 weeks) and post-intervention (6 weeks)
  Wrist-worn actigraphy devices were used to calculate child's 24-hour sleep duration
Child sleep: sleep quality | Baseline (0 weeks) and post-intervention (6 weeks)
  Wrist-worn actigraphy devices were used to calculate child's sleep quality (e.g., wake after sleep onset)
Child sleep: sleep timing | Baseline (0 weeks) and post-intervention (6 weeks)
  Wrist-worn actigraphy devices were used to calculate variability in child's sleep timing

CONTACTS AND LOCATIONS:
Locations (1):
- South Carolina early childhood support state agencies, Columbia, South Carolina, United States